CLINICAL TRIAL: NCT03153267
Title: Duration of Doxycycline Treatment in Patients With Erythema Migrans (EM). A Randomized Clinical Trial.
Brief Title: Duration of Doxycycline Treatment in EM Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: University of Ljubljana School of Medicine, Slovenia (Other)
Responsible Party: Principal Investigator, Daša Stupica, MD, PhD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EM-Doxy714
Record Dates: First submitted 2017-03-16; First posted 2017-05-15 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2019-04

CONDITIONS: Erythema Chronicum Migrans
MeSH Terms: conditions — Erythema Chronicum Migrans | interventions — Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- EM-7 days doxycycline (Active Comparator)
  Interventions: Drug: Doxycycline 100 MG Oral Tablet bid, 7 days
- EM-14 days doxycycline (Active Comparator)
  Interventions: Drug: Doxycycline 100 MG Oral Tablet bid, 14 days
- Controls (Placebo Comparator)
  Interventions: Drug: Controls without a history of lyme disease.

INTERVENTIONS:
Drug: Doxycycline 100 MG Oral Tablet bid, 7 days — Patients will receive doxycycline for 7 days.
  Arms: EM-7 days doxycycline
Drug: Doxycycline 100 MG Oral Tablet bid, 14 days — Patients will receive doxycycline for 14 days.
  Arms: EM-14 days doxycycline
Drug: Controls without a history of lyme disease. — No intervention.
  Arms: Controls

SUMMARY:
The purpose of this study is to compare the efficacy of 7-day versus 14-day doxycycline treatment in patients with erythema migrans.

ELIGIBILITY:
Inclusion Criteria:

* solitary erythema migrans

Exclusion Criteria:

* pregnancy or lactation
* immunocompromised
* serious adverse event to doxycycline
* taking antibiotic with antiborrelial activity within 10 days
* multiple erythema migrans or extracutaneous manifestations of lyme borreliosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Treatment outcome in patients treated for erythema migrans with doxycycline for 7 or 14 days | At 12 months after enrollment.
  Objective sequelae and post-treatment subjective new or increased symptoms (NOIS) in patients treated for erythema migrans with doxycycline for 7 or 14 days.

SECONDARY OUTCOMES:
Comparison of nonspecific symptoms in patients with erythema migrans and control subjects | At 12 months after enrollment.
  Number of patients after treatment with doxycycline for 7 or 14 days for erythema migrans and number of control subjects (without a history o Lyme borreliosis) with nonspecific symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Daša Stupica, MD PhD, Principal Investigator — University Mecical Centre Ljubljana
Locations (1):
- University Medical centzer Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stupica D, Collinet-Adler S, Blagus R, Gomiscek A, Cerar Kisek T, Ruzic-Sabljic E, Veluscek M. Treatment of erythema migrans with doxycycline for 7 days versus 14 days in Slovenia: a randomised open-label non-inferiority trial. Lancet Infect Dis. 2023 Mar;23(3):371-379. doi: 10.1016/S1473-3099(22)00528-X. Epub 2022 Oct 6. PMID 36209759